CLINICAL TRIAL: NCT04101565
Title: Feasibility, Acceptability, & Preliminary Efficacy of Text4Father for Improving Infant & Family Health
Brief Title: Text4Father Pilot Feasibility, Acceptability Study
Acronym: Text4Father
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00226367; 1R21HD097453-01A1 (NIH)
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Fathers; Mhealth; Mobile Health; Nuclear Family
Keywords: Fatherhood

STUDY DESIGN:
Intervention Model Description: 2 groups will be enrolled and randomized to receipt or not receipt of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text4Father (Experimental): Receipt of twice-weekly texts that include resource links and instructions to support behavior change (e.g., videos, infographics) and start mid-pregnancy and continuing through 2 months of baby's age.
  Interventions: Behavioral: Text4Father
- Usual care (No Intervention): Usual care that is consistent with typical maternity care in involving expectant fathers.

INTERVENTIONS:
Behavioral: Text4Father — Receipt of twice-weekly texts that include resource links and instructions to support behavior change (e.g., videos, infographics) and start mid-pregnancy and continuing through 2 months of age.
  Arms: Text4Father

SUMMARY:
This study evaluates the feasibility, acceptability, and preliminary efficacy of Text4Father among first-time lower income fathers. Half of the participants will receive Text4Father - a text messaging educational program - from mid-pregnancy through 2 months of postnatal age, while the other half will receive usual care.

DETAILED DESCRIPTION:
Text4Father, a multi-modal text messaging program, is designed to increase first-time lower income fathers' knowledge, self-efficacy, and behavioral engagement on infant care and parenting. Text4Father consists of 48-weeks of twice weekly texts written at a 5th grade reading level. Texts include resource links and instructions to support behavior change (e.g., videos, infographics), starting mid-pregnancy and continuing through 2 months of postnatal age. Text content was developed using formative research and feedback from the target population, consensus building with experts, and an evidence-based review.

Usual maternity care does not involve expectant fathers in education. Further, while father engagement is widely advocated, few public health and clinical approaches aim to engage expectant fathers during the prenatal period and first months after birth - a critical window of opportunity that has been insufficiently leveraged to promote father engagement when fathers describe being unsure of father role.

ELIGIBILITY:
Inclusion Criteria:

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Self-reported expectant father and pregnant partner (expectant mother)
* Aged ≥18 years
* In a romantic relationship and expect to continue to be in this relationship during the study period
* Able to speak English
* Lower socioeconomic status (SES) (e.g., high school/general education or vocational/trade school or less; or qualify for Medicaid/public insurance, WIC, SNAP, food stamps)
* Access to necessary resources for participating in a technology-based intervention (i.e., cell phone) and willing/able to receive/send texts

Exclusion Criteria:

* Individuals who are not able to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-12-26 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arik V Marcell, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The final version of collected data will be made available within thirty (30) months after the end of the data collection. Data will be preserved and made accessible along with relevant documentation via the chosen repository (e.g., through open access (Open Inter-university Consortium for Political and Social Research (ICPSR)) if possible). Johns Hopkins University School of Medicine will review the disclosure protection of the de-identified datasets. If they conclude that the risk of disclosure is too great for public access, then ICPSR's Traditional Restricted Data or Physical Data Enclave will be used for some or all of the data, with restricted access solely to approved researchers.

REFERENCES:
- [Background] Marcell AV, Johnson SB, Nelson T, Labrique AB, Eck KV, Skelton S, Aqil A, Gibson D. Protocol for the Feasibility, Acceptability, and Preliminary Efficacy Trial of text4FATHER for Improving Underserved Fathers' Involvement in Infant Care. J Health Care Poor Underserved. 2021;32(3):1110-1135. doi: 10.1353/hpu.2021.0117. PMID 34421016
- [Background] Allport BS, Johnson S, Aqil A, Labrique AB, Nelson T, Kc A, Carabas Y, Marcell AV. Promoting Father Involvement for Child and Family Health. Acad Pediatr. 2018 Sep-Oct;18(7):746-753. doi: 10.1016/j.acap.2018.03.011. Epub 2018 Apr 10. PMID 29653255
- [Background] Allport-Altillo BS, Aqil AR, Nelson T, Johnson SB, Labrique AB, Carabas Y, Marcell AV. Parents' Perspectives on Supporting Father Involvement in African American Families During Pregnancy and Early Infancy. J Natl Med Assoc. 2020 Aug;112(4):344-361. doi: 10.1016/j.jnma.2020.04.002. Epub 2020 May 11. PMID 32409095
- [Background] Aqil A, Allport BS, Johnson SB, Nelson T, Labrique AB, Marcell AV. Content to share with expectant fathers: Views of professionals focused on father involvement. Midwifery. 2019 Mar;70:119-126. doi: 10.1016/j.midw.2018.12.018. Epub 2018 Dec 24. PMID 30611921

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 120 participants completed consent procedures, and a total of 97 completed baseline study survey procedures and then were randomized (23 participants did not complete the baseline survey study activity, and were thus not randomized).
Period: Overall Study
Arm/Group | text4FATHER | Usual Care
Started | 53 | 44
Completed | 41 | 34
Not Completed | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | text4FATHER | Usual Care | Total
Number analyzed (Participants) | 53 | 44 | 97
Age, Customized [Count of Participants; unit: Participants]
  18-29 | 33 | 25 | 58
  30 or older | 20 | 19 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 53 | 44 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  non-Hispanic Black | 37 | 30 | 67
  non-Hispanic White | 12 | 11 | 23
  Hispanic | 3 | 2 | 5
  Other | 1 | 1 | 2
Live with partner [Count of Participants; unit: Participants] | 43 | 39 | 82
First-time father [Count of Participants; unit: Participants] | 28 | 16 | 44

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Overall Recruitment
Description: Feasibility of recruitment will be measured as the number of fathers who were randomized and completed baseline procedures.
Time Frame: At Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | text4FATHER | Usual Care
Number analyzed (Participants) | 53 | 44
Participants | 53 | 44

2. Primary Outcome: Feasibility of Overall Retention
Description: Feasibility of retention will be assessed as the number of enrolled participants who complete 7-month follow-up survey (2-months of postnatal age).
Time Frame: Follow-up (7 months)
Measure: Count of Participants; unit: Participants
Arm/Group | text4FATHER | Usual Care
Number analyzed (Participants) | 53 | 44
Participants | 41 | 34

3. Primary Outcome: Intervention Usability as Assessed by the Usability Score
Description: 11 item self-report measure among participating intervention fathers with higher score indicating greater perceived usability of technology (text messaging program). This measure is scaled with range from 1 (low) to 4 (high). Mean of participant scale choice (1-4) is reported.
Time Frame: Follow-up (7 months)
Population: 12 individuals were lost to follow-up & 1 individual did not complete these items
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | text4FATHER
Number analyzed (Participants) | 40
score on a scale | 3.38 (0.39)

4. Primary Outcome: Intervention Acceptability as Assessed by the Acceptability Score
Description: An 9 item self-report measure among participating intervention fathers with higher score indicating greater perceived acceptability of technology (text messaging program). This measure is scaled with range from 1 (low) to 4 (high). Mean of participant scale choice (1-4) is reported.
Time Frame: Follow-up (7 months)
Population: 12 individuals were lost to follow-up & 1 individual did not complete these items
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | text4FATHER
Number analyzed (Participants) | 40
score on a scale | 3.33 (0.51)

5. Secondary Outcome: Self-efficacy as Assessed by the Parenting Sense of Competence Scale (PSOC)
Description: 17 item self-report measure with higher score indicating greater confidence in overall parenting skills to assess Parenting Sense of Competence (PSOC) at follow-up 7 months later (2 months post-birth). This measure is scaled with range from 1 (low) to 6 (high). Mean of participant scale choice (1-6) is reported.
Time Frame: 7 months (2 months post-birth)
Population: 12 intervention fathers were lost to follow-up; 10 usual care fathers were lost to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | text4FATHER | Usual Care
Number analyzed (Participants) | 41 | 34
score on a scale | 4.49 (0.79) | 4.49 (0.60)

ADVERSE EVENTS:
Time Frame: Up to 7 months
Arm/Group | text4FATHER | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/44
Other Adverse Events (participants affected / at risk) | 0/53 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT04101565/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT04101565/ICF_001.pdf